CLINICAL TRIAL: NCT04721548
Title: A Randomized, Double Blind, Parallel-group Study to Evaluate the Efficacy and Safety of a New Pharmaceutical Form Minoxidil 5% for the Treatment of Androgenetic Alopecia in Men for 24 Weeks
Brief Title: Treatment of Androgenetic Alopecia in Men for 24 Weeks
Acronym: MINOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EF171
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at a 2: 1 ratio to receive new pharmaceutical form Minoxidil 5% and placebo, respectively. The primary objective of the MINOX study is to demonstrate the superiority of a new topical 5% pharmaceutical form of minoxidil (experimental drug) in treating men with androgenetic alopecia (Hamilton-Norwood scale IIIv, IV or V) compared to placebo when administered for 180 days.
Who Masked: Participant, Investigator
Masking Description: Masking will be adopted in this study, in which the experimental products under evaluation will be provided in a masked way, that is, one group will receive an experimental drug (Minoxidil 5%) and another group will receive a placebo (product without the active ingredient) in identical primary and secondary packaging to avoid potential bias, so neither the researcher nor the research participant will know what is being applied.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minoxidil´s Placebo (Placebo Comparator): The recommended dosage is 1 ml of the solution twice a day (morning and evening).
  Interventions: Drug: Placebo
- Topical Minoxidil 5% (Experimental): The recommended dosage is 1 ml of the solution twice a day (morning and evening).
  Interventions: Drug: Minoxidil Topical Foam

INTERVENTIONS:
Drug: Minoxidil Topical Foam — Apply 1 mL of solution twice a day.
  Arms: Topical Minoxidil 5%
Drug: Placebo — 1 mL of solution twice a day.
  Arms: Minoxidil´s Placebo

SUMMARY:
A prospective, randomized, double-blind, single-center, placebo-Controlled, parallel-group study to evaluate the efficacy and safety of a new pharmaceutical form Minoxidil 5% in men after 24 weeks of treatment.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
Participants will be randomized at a 2: 1 ratio to receive new pharmaceutical form Minoxidil 5% and placebo, respectively. Through this method, it is possible to obtain more information about the effectiveness of investigational product.

The primary objective of the MINOX study is to demonstrate the superiority of a new topical 5% pharmaceutical form of minoxidil (experimental drug) in treating men with androgenetic alopecia (Hamilton-Norwood scale IIIv, IV or V) compared to placebo when administered for 180 days.

Secondary objectives: 1- To evaluate the efficacy of a new topical 5% minoxidil pharmaceutical form in the treatment of men with androgenetic alopecia, compared to placebo, by means of terminal strand density in the target area, evaluated 30 (±3), 60(±3), 90(±3) and 135(±3) days after the beginning of treatment.

2- To evaluate the efficacy of a new topical 5% pharmaceutical form of minoxidil in the treatment of men with androgenetic alopecia, compared to placebo, by means of the percentage of anagen strands in the target area, evaluated 30(±3), 60(±3), 90(±3), 135(±3) and 180(±3) days after the start of treatment.

3- Evaluate the efficacy of a new topical 5% pharmaceutical form of minoxidil in the treatment of men with androgenetic alopecia, compared to placebo, by means of the average length of hair strands in the target area, evaluated 30(±3), 60(±3), 90(±3), 135(±3) and 180(±3) days after the start of treatment.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years;
* Male pattern baldness identified according the Norwood Hamilton scale: stage IIIv vertex, stage IV, or stage V;
* Terminal hair density equal to or less than 220 hairs/cm2 measured with the Trichoscale Al;
* Subjects who are willing and able to comply with all requirements of the study for the intended period;
* Subjects who give their consent to the study after thoroughly clarification and who personally signed and dated the informed consent document has been informed of all pertinent aspects of the trial;

Exclusion Criteria:

* Current or 6 months dated back use of:
* Minoxidil, finasteride, or any 5 alpha-reductase inhibitor;
* Medications that can potentiate Hypertrichosis, such as: cyclosporine, phenytoin, psolarenes, oral glucocorticoids (except inhalers), lithium, phenothiazinics
* Medications with anti-androgenic properties, such as: cyproterone, spironolactone, ketoconazole, flutamide, bicalutamide.
* Any anabolic steroid ;
* Current or 8 weeks dated back use of herbal products such as saw palmetto;
* Isotretinoin for at least 12 months;
* Current or 2 weeks dated back use of dietary or vitamin supplements;
* Subjects who had a dignosis of malignant disease in the alopecia area in the period of 05 years;

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 336 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Absolute change in terminal thread density in the target area determined 180 (±3) days after the start of treatment compared to baseline density. | 24 weeks
  The density of terminal hairs will be evaluated by phototrichogram (FotoFinder leviacam® and Trichoscale Al® Dermatoscope), with the baseline density resulting from the images captured on the VR and VR+2 days visits and the final density resulting from the images captured on the V5 and V5+2 days visits. Terminal wires will be classified as those with diameter greater than or equal to 30 um.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No